CLINICAL TRIAL: NCT03914781
Title: Feasibility Trial of an Internet-based Self-management Program to Improve Disease-management Self-efficacy in Patients With Scleroderma: A Scleroderma Patient-centered Intervention Network (SPIN) Study
Brief Title: SPIN Self-Management Feasibility Trial
Acronym: SPIN-SELF-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Senior Investigator, Lady Davis Institute for Medical Research, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-1146
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Scleroderma; Systemic Sclerosis; Self-management; E-health; Intervention
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIN-SELF program (Experimental): Offered access to the online SPIN-SELF program in addition to usual care
  Interventions: Behavioral: SPIN-SELF Program
- Not Offered the SPIN-SELF program (No Intervention): Usual care

INTERVENTIONS:
Behavioral: SPIN-SELF Program — The SPIN-SELF program utilizes social modelling through educational videos of scleroderma patients who describe their own challenges and what they have done to cope with living with scleroderma, as well as videos of patients and health professionals who teach key self-management techniques. The program includes sections on general self-management skills, including goal-setting and self-monitoring), progress tracking, sharing goals and progress with friends and family, and patient stories of experiences with using self-management techniques to cope with SSc symptoms. The program's 9 modules focus on (1) coping with pain; (2) skin care, finger ulcers and Raynaud's; (3) sleep problems; (4) fatigue; (5) gastrointestinal symptoms; (6) itch; (7) managing emotions and stress; (8) coping with body image concerns due to disfigurement; and (9) effective communication with healthcare providers.
  Arms: SPIN-SELF program

SUMMARY:
The Scleroderma Patient-centered Intervention Network (SPIN) is an organization established by researchers, health care providers, and people living with scleroderma (systemic sclerosis; SSc) from Canada, the United States, Mexico, Australia, France, Spain, and the United Kingdom. The objectives of SPIN are (1) to assemble a large cohort of SSc patients who complete outcome assessments regularly in order to learn more about important problems faced by people living with SSc and (2) to develop and test a series of internet-based interventions to help patients manage problems related to SSc, including a self-management program (SPIN-SELF Program).

In the SPIN-SELF feasibility trial, eligible SPIN Cohort participants will be randomized to be offered the SPIN-SELF Program (in addition to usual care) or to usual care only. The SPIN-SELF Program was designed by SPIN members based on key tenets of behaviour change that have been successfully incorporated in programs for more common diseases and on patient input. It utilizes social modelling through educational videos of SSc patients describing their challenges and what they have done to cope with SSc, as well as videos teaching key self-management techniques. After an introduction to self-management and instructions on how to navigate the program, a short quiz comprised of one-item questions will direct patients to modules that are most relevant to their symptoms and disease management challenges. The program's modules address (1) pain; (2) skin care, finger ulcers, and Raynaud's; (3) sleep problems; (4) fatigue; (5) gastrointestinal symptoms; (6) itch; (7) emotions and stress; (8) body image concerns due to disfigurement; and (9) effective communication with healthcare providers.

The aim of the SPIN-SELF feasibility study is to collect data to assess the feasibility of planned procedures for the full-scale trial; required resources; and scientific aspects of the study (e.g., withdrawal rate, outcomes measures). These data will be used to determine whether it is feasible to carry out the main trial or whether changes need to be made before conducting a full-scale RCT of the SPIN-SELF Program.

DETAILED DESCRIPTION:
The SPIN Cohort currently includes over 1800 SSc patients from 41 sites in Canada, the United States, Mexico, Australia, and France, Spain, and the United Kingdom. SPIN Cohort participants complete outcome measures via the Internet upon enrolment and subsequently every three months. SPIN utilizes the cohort multiple RCT (cmRCT) design as a framework for conducting trials of interventions. SPIN Cohort participants consent to allow personal data to be used for observational research, to assess intervention trial eligibility and, if eligible, to be randomized. Participants also consent that, if eligible and randomized to usual care, the participants' data can be used to evaluate intervention effectiveness without the participants being notified that they have been randomized to the usual care group and not offered the intervention. Thus, in SPIN trials, trial status is masked for participants in the control arm, who are not aware that they are participating in the trial, but not for participants in the intervention arm. The investigative team does not interact with patients for care provision or outcome assessment, which are done automatically via the internet.

The SPIN-SELF feasibility study is embedded in the SPIN Cohort and will evaluate the feasibility of conducting a full-scale RCT of the SPIN-SELF Program. Investigators will randomize 40 SPIN Cohort participants with low disease management self-efficacy and an indicated interest in using an online self-management program to be offered the SPIN-SELF Program or usual care only.

Randomization will occur at the time of participants' regular SPIN Cohort assessments. Eligible participants, based on questionnaire responses, will be randomized automatically using simple 3:2 randomization, using a feature in the SPIN Cohort platform, which provides immediate randomization and complete allocation sequence concealment.

Feasibility outcomes include participant eligibility and recruitment, and numbers and percentages of participants who do not respond to follow-up measures. Use of the online intervention will be described by presenting the frequency of logins and time spent on the SPIN-SELF Program. Analysis of outcome measures will include the completeness of data and presence of floor or ceiling effects. Descriptive statistics will be used to provide means and standard deviations for the measures. Qualitative information and information related to management and usability of the SPIN-SELF Program will inform any necessary changes to the intervention or trial procedures.

ELIGIBILITY:
Inclusion Criteria:

* SPIN Cohort patients must have a systemic sclerosis (SSc) diagnosis based on 2013 American College of Rheumatology/European League Against Rheumatism criteria confirmed by a SPIN physician, be ≥18 years old, be able to give informed consent, and be fluent in English, French or Spanish.
* For the feasibility trial, eligible patients must be able to use the online intervention in English, have low disease management self-efficacy (Self-Efficacy for Managing Chronic Disease (SEMCD) ≤ 7), have indicated high interest in using an online self-management intervention (≥6 on 0-10 scale).

Exclusion Criteria:

* Patients not able to access or respond to questionnaires via the internet are excluded.
* Participants who are currently participating in another SPIN intervention trial and have not yet completed their final assessment measures will be excluded.
* French and Spanish speaking participants will be excluded from the feasibility trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Eligibility: Number of patients in the SPIN Cohort who meet the cut-off thresholds for eligibility | Baseline
  Measure: count of eligible patients
Enrolment: Percentage of patients who consent to participation | Baseline
  Measure: count of consenting patients
Participant feedback on usability | 3 months
  Participant interviews
Intervention use: Number of logins and time spent on the SPIN-SELF program | 3 months
  Measure: usage log data
Usage log data: Completeness of the automatic usage log data values collected | 3 months
  Measure: usage log data
Usage log data: Linking of data from the SPIN Cohort and SPIN-SELF platforms | 3 months
  Measure: usage log data
Technological problems | 3 months
  Measure: count of technological problems reported by staff and participants

SECONDARY OUTCOMES:
Self-Efficacy for Managing Chronic Disease (SEMCD) Scale | Baseline, 3 months
  The 6-item SEMCD Scale measures self-efficacy among patients with chronic medical conditions by asking them to rate their confidence that they can perform certain tasks related to managing their disease. Items are rated on a numerical scale ranging from 1 (not confident at all) to 10 (totally confident). The score for the scale is the mean of all item scores, with higher scores reflecting greater self-efficacy
Patient Reported Outcomes Measurement Information System (PROMIS-29) profile version 2.0 | Baseline, 3 months
  Measures 8 domains of health status with 4 items for each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference) plus a single item for pain intensity. Items are scored on a 5-point scale (range 1-5), with different response options for different domains, and the single pain intensity item is measured on an 11-point rating scale. Higher scores represent more of the domain being measured

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request

REFERENCES:
- [Derived] Kwakkenbos L, Ostbo N, Carrier ME, Nielson WR, Fedoruk C, Levis B, Henry RS, Pope J, Frech T, Gholizadeh S, Johnson SR, Piotrowski P, Jewett LR, Gordon J, Chung L, Bilsker D, Tao L, Turner KA, Cumin J, Welling J, Fortune C, Leite C, Gottesman K, Sauve M, Reyna TSR, Hudson M, Larche M, van Breda W, Suarez-Almazor ME, Bartlett SJ, Malcarne VL, Mayes MD, Boutron I, Mouthon L, Benedetti A, Thombs BD; SPIN Investigators. Randomized feasibility trial of the Scleroderma Patient-centered Intervention Network Self-Management (SPIN-SELF) Program. Pilot Feasibility Stud. 2022 Feb 26;8(1):45. doi: 10.1186/s40814-022-00994-5. PMID 35219340